CLINICAL TRIAL: NCT03915093
Title: Thoracoscopic Surgery: Effect of Designing and Implementing Educational Nursing Protocol on Patients Quality of Life
Brief Title: Effect of Prehabilitation Protocol on Quality of Life After Thoracoscopic Surgery
Acronym: VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Nafady Abd El Hafez, Assisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1562017
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Thoracoscopy; Prehabilitation
Keywords: Thoracoscopy; Educational nursing protocol; Quality of life

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): receive educational nursing protocol
  Interventions: Other: Educational nursing protocol; Other: Routine hospital care
- control group (Active Comparator): receive routine hospital care
  Interventions: Other: Routine hospital care

INTERVENTIONS:
Other: Educational nursing protocol — It is a booklet given to study group ,which contains Knowledge and practice about thoracoscopy, pre - post operative care and home care instructions
  Arms: study group
Other: Routine hospital care — The routine care given by physicians and nurses after thoracoscopic surgery

SUMMARY:
video-assisted thoracic surgery (VATS) is a new approach used in cardio thoracic surgery department instead of thoracotomy to treat several diseases.patients underwent thoracoscopic surgery without organized educational protocol either before or after the procedure. Therefore, this study will be the first clinical research which will increase patients' knowledge about thoracoscopy and decrease its complications.

DETAILED DESCRIPTION:
The role of thoracic nursing specialty is to support and educate patients, who are suffering from thoracic diseases, to achieve the best outcome in terms of physical, psychological, social and spiritual well beings. The care provided not only focuses on in-hospital treatments that patient received, but also encompasses the whole patient journey including lifestyle modification, health concept promotion, self-empowerment and secondary prevention. Preoperative prophylactic physiotherapy has been shown to be an important and effective approach in preventing or reducing postoperative complications, in addition to optimizing treatment by familiarizing the patient with the physiotherapeutic procedures. Quasi experimental research design was utilized to conduct this study.Sixty adult patients undergoing thoracoscopic surgery included and had the following criteria, the age ranged from 18-65 years old, both male and female. The patients divided into two equal groups (study and control groups), 30 patients for each. The study group received educational nursing protocol while the control group received the routine hospital care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergoing thoracoscopic surgery
* Age 18-65 year
* patients who agree to participate in the study

Exclusion Criteria:

* converting to thoracotomy
* patients refuse to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Effect of prehabilitation on quality of life after thoracoscopic surgery | after one month postoperative
  WHOQOL developed by WHO (2004). It contains 5 broad domains of QOL within which 18 facets are covered to determine the quality of life. These 5 domains include physical, social, psychological, environmental and perceived QOL. Within each domain several sub domains (facets) of QOL Summarize that particular domain of QOL.The scoring of these variables, a 3-point lickert scale on tables was adopted for the answer low QOL=0-3, moderate QOL=4-6, and high QOL =7-9.

SECONDARY OUTCOMES:
effect of prehabilitation on duration of hospital stay after thoracoscopic surgery | immediate post operative
  assess length of hospital stay postoperative for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Hussein El Khayat, Study Director — faculty of medicine; Sahra Azer, Study Director — faculty of nursing; Magda Mohamed, Study Director — faculty of nursing
Locations (1):
- Assiut U, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeung WW. Post-operative care to promote recovery for thoracic surgical patients: a nursing perspective. J Thorac Dis. 2016 Feb;8(Suppl 1):S71-7. doi: 10.3978/j.issn.2072-1439.2015.10.68. PMID 26941973
- [Background] Gao K, Yu PM, Su JH, He CQ, Liu LX, Zhou YB, Pu Q, Che GW. Cardiopulmonary exercise testing screening and pre-operative pulmonary rehabilitation reduce postoperative complications and improve fast-track recovery after lung cancer surgery: A study for 342 cases. Thorac Cancer. 2015 Jul;6(4):443-9. doi: 10.1111/1759-7714.12199. Epub 2014 Dec 22. PMID 26273399